CLINICAL TRIAL: NCT03756337
Title: Comparison of Audiometric Performance Between the Neuro 1 and Neuro 2 Sound Processors.
Brief Title: Neuro 1 vs. Neuro 2 Sound Processors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PIC-20
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Hearing Loss, Sensorineural; Cochlear Hearing Loss
Keywords: cochlear implant; sound processor; upgrade
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro 2 Upgrade (Experimental): Participant wears Neuro 1 sound processor and is tested, then is upgraded with the new sound processor Neuro 2 and tested.
  Interventions: Device: Neuro 1 & Neuro 2
- Neuro 1 Downgrade (Experimental): Participant wears Neuro 2 sound processor and is tested, then is downgraded with the sound processor Neuro 1 and tested.
  Interventions: Device: Neuro 2 & Neuro 1

INTERVENTIONS:
Device: Neuro 1 & Neuro 2 — participant common fitting map used for tests
  Arms: Neuro 2 Upgrade
Device: Neuro 2 & Neuro 1 — participant common fitting map used for tests
  Arms: Neuro 1 Downgrade

SUMMARY:
This study evaluates the benefit of Neuro 1 sound processor upgrade in speech perfomance in adults. Half of participants will be tested with Neuro 1 first and Neuro 2, while the other half will be tested with Neuro 2 first and then Neuro 1.

DETAILED DESCRIPTION:
The Neuro 1 processor represented a technological advancement over past models, particularly in detecting the environment and automatically adjusting to the sound environment. A second version of the Neuro 1 processor has been developed, the Neuro 2. The signal processing and stimulation characteristics are similar, so speech comprehension levels are expected to be equivalent. This study is designed to compare Neuro 1 and Neuro 2 in terms of audiometric performance.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* primary implantation
* subject having participated to previous Neuro 1 sound processor study in Canada
* fluent in English, including reading and writing.

Exclusion Criteria:

* psychologically unsuitable
* unrealistic expectations regarding possible benefits, risks, and limitations that are inherent to the device
* non compliant with all investigational requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
speech recognition in quiet | Day 1
  Hearing In Noise Test

SECONDARY OUTCOMES:
speech recognition in noise | Day 1
  Hearing In Noise Test
pure tone threshold | Day 1
  from 250Hz to 8kHz

CONTACTS AND LOCATIONS:
Overall Officials: David Peter Morris, MD, Principal Investigator — Dalhousie University, Halifax,NS, Canada
Locations (1):
- Nova Scotia Hearing and Speech centres, Halifax, Canada

IPD SHARING:
Plan to Share IPD: No